CLINICAL TRIAL: NCT04406415
Title: A Single-Center, Double-Blind, Placebo-Controlled, Phase 1b Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Sequential Dose Regimens of Oral Nafamostat Mesylate in Healthy Volunteers Subjects
Brief Title: Oral Nafamostat in Healthy Volunteers (NAF-101)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NAF-101; UG3DA047682-02 (NIH)
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — nafamostat

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, Multiple Ascending Dose (MAD) study with 4 active drug cohorts
Who Masked: Participant
Masking Description: This is a double-blinded study. Subjects will not be informed of their treatment assignment (active or placebo); however, investigators and clinical site staff will have access to the randomization codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- 10 mg (Experimental): 10 mg nafamostat three times a day (t.i.d., approximately q8h) for up to 5 days
  Interventions: Drug: Nafamostat Mesilate
- 50 mg (Experimental): 50 mg nafamostat three times a day (t.i.d., approximately q8h) for up to 5 days
  Interventions: Drug: Nafamostat Mesilate
- 100 mg (Experimental): 100 mg nafamostat three times a day (t.i.d., approximately q8h) for up to 5 days
  Interventions: Drug: Nafamostat Mesilate
- 200 mg (Experimental): 200 mg nafamostat three times a day (t.i.d., approximately q8h) for up to 5 days
  Interventions: Drug: Nafamostat Mesilate
- Placebo (Placebo Comparator): Placebo administered three times a day (t.i.d., approximately q8h) for up to 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nafamostat Mesilate — Oral nafamostat, 10, 50, 100, or 200 mg administered three times daily for up to 5 days
  Arms: 10 mg; 100 mg; 200 mg; 50 mg
Drug: Placebo — Oral placebo administered three times daily for up to 5 days
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Multiple Ascending Dose (MAD) study to evaluate the safety, tolerability and pharmacokinetics of oral nafamostat solution administered t.i.d.. for up to 5 days in healthy volunteer adult subjects

DETAILED DESCRIPTION:
Subjects will undergo a medical screening (Days -1 to -10) and, if eligible, informed consent will be obtained prior to 6 days of confinement at the clinic site. Up to 20 subjects will be randomized. Subjects will be stratified to include an equal number of male and female subjects who will receive active drug within each dose cohort, and an equal number of male and female subjects in the combined placebo group. Separate groups of volunteers will be used for each dose cohort. There will be 4 dose cohorts in this study with active drug doses of 10, 50, 100, and 200 mg nafamostat in succeeding cohorts. Each cohort of 5 subjects will enroll 2 male and 2 female to receive active drug and 1 subject (male or female) to receive placebo for a total of 20 subjects. The placebo subject from each cohort will be combined into a placebo cohort that will have 4 subjects to compare to 4 subjects in each of the active dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 to 70 years old, able and willing to provide written informed consent to participate in the study;
2. Subjects must be in generally good health as determined by pre-study medical history, physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG);
3. Subjects must be willing to remain in confinement at the clinical study unit for 6.5 consecutive days and to return to the unit at Day 14±2 for followup safety assessments;
4. Body mass index (BMI) 19-32 kg/m2;
5. Normal blood pressure (BP) [systolic BP 90-140 mmHg, diastolic BP 50-90 mmHg] and heart rate (HR) [resting HR 45-90 beats per minute (bpm)] without medication;
6. Clinical chemistry profile including electrolytes, alkaline phosphatase (ALK), lactate dehydrogenase (LDH), creatine phosphokinase (CPK), creatinine, and urea must be within the normal range without medication; screening liver enzymes may be up to 1.5x normal range; screening CPK must be within 2x normal range;
7. Urinalysis including urinary creatinine must be within normal limits (trace findings and minor deviations are acceptable per the clinical decision of the Principal Investigator);
8. Subjects must be non-smokers or willing to abstain from smoking for the duration of study;
9. Subjects must be able to read, understand and follow the study instructions;
10. Male subjects and their female sexual partners must agree to use double barrier contraception during the study period and for 2 months afterward, or provide proof of post-menopausal state (minimum 1 year) or surgical sterility.
11. Female subjects will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, or surgically sterile for at least 3 months, or will agree to use double-barrier contraception from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 2 months after Clinic Discharge. Double barrier contraception may include, but is not limited to, non-hormonal intrauterine device with spermicide, female condom with spermicide, diaphragm with spermicide, cervical cap with spermicide; having a male sexual partner who agrees to use a male condom with spermicide; or having a sterile sexual partner. Females will refrain from using hormonal contraceptives for at least 28 days prior to study entry until the end of the study period (Day 14). For all females, the pregnancy test result must be negative at Screening and Pre-Study Baseline (Days -1 to -10).

Exclusion Criteria:

1. Use of any non-study medication(s) including low dose aspirin for cardiovascular prophylaxis within one week prior and two weeks after receipt of study drug;
2. Use of chemotherapy agents or history of cancer, other than non-metastatic skin cancer that has been completely excised, within five years prior to the screening visit;
3. History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 1 month of study;
4. History of congestive heart failure;
5. Use of drugs which are P450 inducers or inhibitors within the past 30 days (e.g. cimetidine, paroxetine, fluoxetine, haloperidol, ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin);
6. Use of any dietary aids or foods that are known to modulate drug metabolizing enzymes (e.g. St. John's Wort, grapefruit juice) within 14 days of dose administration;
7. History of seizure disorder;
8. Serious psychosocial co-morbidities;
9. Cognitive or psychiatric disorders, or any other condition that could interfere with compliance with study procedures and/or confinement in a clinical study unit for 6.5 days;
10. History of drug or alcohol abuse within one year prior to screening;
11. Use of any other investigational drug within 1 month prior to enrollment;
12. Use of prescription drugs within 1 month prior to enrollment;
13. Use of over the counter medication excluding routine vitamins, but including mega-dose vitamin therapy, within one week of enrollment;
14. Donation and/or receipt of any blood or blood products within 3 months prior to enrollment;
15. Family history of significant cardiac disease (i.e. sudden death in first degree relative; myocardial infarction prior to 50 years old).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 14 Days
  Number of participants with adverse events including out-of-range clinical laboratory measures, vital signs, ECG, and spontaneous adverse event reports throughout the 14 day study period

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Pre-dose (0 hr) and at 0.5, 1, 2, 3, 4, 6, and 8 hr after first dose on Day 1 and again after the last dose on Day 5
  Peak plasma concentrations of nafamostat
Pharmacokinetics (Tmax) | Pre-dose (0 hr) and at 0.5, 1, 2, 3, 4, 6, and 8 hr after first dose on Day 1 and again after the last dose on Day 5
  Time to peak plasma concentrations of nafamostat
Pharmacokinetics (AUC) | Pre-dose (0 hr) and at 0.5, 1, 2, 3, 4, 6, and 8 hr after first dose on Day 1 and again after the last dose on Day 5
  Area under the plasma concentration vs. time curve (AUC) for nafamostat
Dose Selection | 5 Days
  Identify dose of nafamostat to maintain a concentration of 3.5 ng/mL (10 nM) or higher for 4 hours or longer after each dose

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — Ensysce Biosciences
Locations (1):
- Arizona Research Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No